CLINICAL TRIAL: NCT05213221
Title: Study on Therapeutic Effect of Combination of Envafolimab, Lenavatinib and TACE in Advanced HCC Patients: an Open, Single Arm, Phase II Clinical Trial
Brief Title: Study on Therapeutic Effect of Combination of Envafolimab, Lenavatinib and TACE in Advanced HCC Patients
Acronym: CISLD-12
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, The chairman of the First Affiliated Hospital of Zhejiang University School of Medicine, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CISLD-12
Record Dates: First submitted 2021-12-21; First posted 2022-01-28 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Advanced Hepatocellular Carcinoma
MeSH Terms: interventions — envafolimab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Envafolimab, Lenvatinib and TACE
  Interventions: Drug: Envafolimab; Procedure: TACE; Drug: Lenvatinib

INTERVENTIONS:
Drug: Envafolimab — 300mg, subcutaneous injection, q3w
Procedure: TACE — The first TACE will be started on d1, and the subsequent TACE will be performed on demand.
Drug: Lenvatinib — 8mg,QD (body weight <60kg); 12mg, QD (body weight ≥ 60kg)

SUMMARY:
This study is a single-center, open, single-arm, phase II clinical trial. Eligible HCC patients, after signing informed consent, will receive TACE treatment. Envafolimab combined with Lenvatinib will be started on the day of TACE, and the subsequent TACE will be performed on demand. Patients will receive the treatment continuously until disease progression or intolerance. Tumor imaging evaluation will be performed according to RECIST V1.1 criteria every 6 weeks. Safety will be assessed with CTCAE 5.0. Adverse events throughout and within 30 days of the end of the study will be recorded (severe adverse events or adverse events associated with Envafolimab will be recorded within 90 days after the end of treatment).Treatment will last for 2 years or until disease progression, withdrawal of informed consent, loss of visit, or death.

ELIGIBILITY:
Inclusion Criteria:

* Sign a written informed consent form prior to enrollment;
* Age was 18-75 years old;
* Hepatocellular carcinoma (HCC) was confirmed by imaging or histology or cytology;
* Patients with stage C and B unresectable BCLC stage (either with portal cancer emboli including VP1-3, but not enrolled if the main portal cancer embolus completely blocked blood vessels and had no blood flow passage)
* With measurable foci (non-lymph node lesion CT scan long diameter ≥ 10 mm, lymph node lesion CT scan short diameter ≥ 15 mm according to RECIST 1.1 criteria);
* Has never previously received any antitumor system treatment, especially the immunotherapy;
* ECOG score: 0~1;
* Child-Pugh score ≤ 7;
* Have adequate organ function;
* Estimated survival period of ≥ for 3 months;

Exclusion Criteria:

* Previously diagnosed by histology/cytology with fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma and other components.
* The patient has suffered from other malignant tumors in the past or at the same time.
* Patients who have received systemic anti-tumor therapy in the past;
* For HCC lesions ≥10cm in any dimension, there are more than 10 lesions evaluated by imaging or HCC lesions account for ≥50% of the liver volume;
* Is a current candidate for liver transplantation or has experienced liver transplantation;
* There is a risk of bleeding, or coagulation dysfunction, or is undergoing thrombolytic therapy; or has had bleeding from esophageal or gastric varices in the past 6 months;
* Portal vein tumor thrombus Vp4.
* The patient is known to have been allergic to macromolecular protein preparations or applied drug components;
* The patient has any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis Patients with abnormal thyroid function (hyperthyroidism/decreased thyroid function), and the use of drugs cannot maintain thyroid function in the normal range, or previous thyroid surgery, patients who need long-term thyroxine and other drug replacement therapy after surgery; the patient has Vitiligo or asthma has been completely relieved in childhood, and those without any intervention after adulthood can be included; asthma whose patients require medical intervention with bronchodilators cannot be included)
* The patient is using immunosuppressive agents, or systemic or absorbable local hormone therapy to achieve immunosuppressive purposes (dose>10mg/day prednisone or other curative hormones), and within 2 weeks before enrollment Still in use;
* The patient is still using traditional Chinese medicine or other immunomodulators within 2 weeks before enrollment;
* Ascites or pleural effusion with clinical symptoms cannot be controlled with drugs and requires therapeutic puncture or drainage;
* There are clinical symptoms or diseases of the heart that are not well controlled, such as: (1) Heart failure above NYHA level 2 (2) Unstable angina (3) Myocardial infarction occurred within 1 year (4) Supraventricular with clinical significance Or patients with ventricular arrhythmia in need of treatment or intervention;
* Severe infections that are active or poorly clinically controlled. Severe infections within 4 weeks before the first administration, including but not limited to hospitalization due to complications of infection, bacteremia or severe pneumonia, or fever of unexplained occurrence> 38.5 degrees during the screening period and before the first administration (by research According to the judge, the patient can be included in the group for fever caused by the tumor);
* Past and current patients with objective evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, severely impaired lung function, etc.; patients with known syphilis infection requiring treatment; active tuberculosis ( Active tuberculosis, TB), who are receiving anti-tuberculosis treatment or have received anti-tuberculosis treatment within 1 year before the first administration.
* patients with congenital or acquired immune deficiencies, such as HIV infection, or active hepatitis (transaminase does not meet the selection criteria, hepatitis B reference: HBV DNA ≥2000 IU/ml or ≥104 copies/ml; hepatitis C reference: HCV RNA≥2000 IU/ml or ≥104 copies/ml; after nucleotide antiviral therapy, it is lower than the above standard and can be included in the group); chronic hepatitis B virus carriers, HBV DNA<2000 IU/ml, test During this period, you must receive antiviral treatment at the same time before you can join the group;
* Live vaccines may be vaccinated during the study period less than 4 weeks before the study medication;
* The patient is known to have a history of psychotropic drug abuse, alcohol abuse or drug abuse;
* The investigator believes that it should be excluded from the study. For example, the investigator judges that the patient has other factors that may cause the study to be terminated halfway, such as other serious diseases (including mental illness) that require combined treatment. Serious laboratory abnormalities, accompanied by family or social factors, can affect the safety of patients or the collection of data and samples.
* The patient has metastases to the central nervous system.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Objective reponse rate (ORR) | Up to 2 years.
  The proportion of patients who had tumor evaluated as PR according to RECIST1.1 criteria during study

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to 2 years.
  The proportion of patients who had tumor evaluated as PR or SD according to RECIST1.1 criteria during study
Duration of remission （DoR） | Up to 2 years.
  The time from the first assessment of the tumor as CR or PR to the first assessment of PD or death from any cause.
Progression-free survival （PFS） | Up to 2 years.
  The time from enrolled to disease pregression or death from any cause.
Overall survival (OS) | Up to 2 years.
  The time from enrolled to death from any cause.
Safety of treatment | Up to 2 years.
  Safety evaluation was done continuously during treatment by using CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Tingbo Liang, PhD, Study Chair — Zhejiang University
Locations (1):
- the First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen Y, Zhang J, Hu W, Li X, Sun K, Shen Y, Zhang M, Wu J, Gao S, Yu J, Que R, Zhang Y, Yang F, Xia W, Zhang A, Tang X, Bai X, Liang T. Envafolimab plus lenvatinib and transcatheter arterial chemoembolization for unresectable hepatocellular carcinoma: a prospective, single-arm, phase II study. Signal Transduct Target Ther. 2024 Oct 9;9(1):280. doi: 10.1038/s41392-024-01991-1. PMID 39384742